CLINICAL TRIAL: NCT03677206
Title: The Effect of Light Therapy on Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Mohab Ibrahim, PhD MD, Director, Comprehensive Pain Management Clinic Associate Professor, Anesthesiology, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1604514512
Record Dates: First submitted 2017-05-11; First posted 2018-09-19 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Initially, patients will receive White LED exposure, then they will be crossed over to Green LED exposure. The patients will not be told which one is the treatment and which one is the control.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exposure to white LED light. (Sham Comparator): Subjects will exposed to white light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks
  Interventions: Device: Exposure to white LED light
- Exposure to green LED light (Experimental): Subjects will exposed to green light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks.
  Interventions: Device: Exposure to green LED light
- Cross over (Other): Subject will be exposed to white light (sham) for 10 weeks, then have a wash out period for 2 weeks, then exposed to green light (experimental) for 10 weeks.
  Interventions: Device: Exposure to green LED light; Device: Exposure to white LED light

INTERVENTIONS:
Device: Exposure to green LED light — Participants will be exposed to green LED strip lights in a dark room for 2 hours a day.
  Arms: Cross over; Exposure to green LED light
Device: Exposure to white LED light — Participants will be exposed to white LED strip lights in a dark room for 2 hours a day.
  Arms: Cross over; Exposure to white LED light.

SUMMARY:
Chronic pain is a major problem in the USA and the rest of the world, currently, all available pharmacological interventions carry with them significant side effects. Pain clinics are specially equipped to perform intentional pain procedures to manage pain. However, there remain groups of patients what neither benefit from pharmacological nor from interventional pain procedures. Other methods have shown only minor benefits such as hypnosis or cognitive behavioral therapy. Therefore, other techniques need to be investigated.

Light therapy has been shown to have significant biological effects on humans. For example, light therapy is used to manage depression. Several clinical trials have shown that certain wavelengths of light can improve wound healing, decrease temporomandibular joint dysfunction (TMJ) pain, and decrease fear of back pain. In these trials, light was directed at the site of pain. In an attempt to better understand the effect of different wavelengths of light, pre-clinical studies were conducted using rats. The investigators have shown green and blue Light emitting diode, (LED) light produced antinociception (analgesia) and reversed neuropathic pain associated with several models of chronic pain. The analgesic effect of light was completely blocked when rats had their eyes covered, this suggests that the analgesic effects seen are mainly due to systemic effect through the visual system.

Preliminary experiments on rats suggest that this effect is mediated through the endogenous opioids and cannabinoid system.

The investigators believe that LED light is a safe alternative to pharmacological intervention to manage pain by stimulating the endogenous endorphin and cannabinoid systems. The investigators initial target participants with history of HIV, chemotherapy induced peripheral neuropathy and fibromyalgia. Participants will be divided into 2 groups. The first group will be a control group exposed to white LED light. The second group will be exposed to green LED light, respectively. Participants will be asked to take LED light home and will be asked to set in a dark room for 2 hours daily for 3 months with their LED light on. At the end of the 3 months trial, the investigator will assess their pain intensity, analgesic use, and overall quality of life. The investigators hypothesis is that participants exposed to green and blue light will have less use of analgesics and will have better life quality.

DETAILED DESCRIPTION:
During the initial visit, the investigator will collect several pieces of data from participants that are considered part of the routine care, if you are being seen in the clinic, this information will also be used for research purposes. Initially the investigator will ask participants to provide their age, gender, work status, disability status, type of work, whether a previous pain physician has evaluated or provided treatment in the past, if there is any ongoing litigation, a detailed description of the pain (burning, electrical, shooting…etc.) and its location. If the participants are being seen in the clinic for their normal care a detailed physical examination assessing the motor strength of the upper extremities, sensation to light touch and reflexes that is part of the standard of care will be provided for the participants. The participants will be asked to give a numerical value for their pain (a scale from 0-10 where 0 is no pain and 10 is the worst pain imagined). Two questionnaires will be provided for the participants to complete which are not standard of care. The first one is the EuroQol Group (EQ-5D) which provide an over assessment of the quality of life. The second is a medication log to document their analgesics use. If the participants are being evaluated via telephone call, the same questions will be conducted, but no physical exam will be provided.

The participants will be assigned to either a white, or green light group. The participants have 50% chance of being in either group. Once the participants are assigned a light group, the participants will be given a strip of Light emitting diode, (LED) light that correspond to their color group. The participants will be asked to take and use the LED strip in a dark room in their house every day for two hours to be exposed to the light, the participants will do this for 10 weeks. The study start date and the outcome assessment timeline will begin from the date of your first exposure to the assigned light. The participants will be asked to complete their weekly questionnaires and daily log, these will be given to the participants on their first clinic visit or sent to the participants if they live out of town. There will be several follow up appointments as detailed below. There is a chance the participants may be asked to cross over into a different group from the one the participants were assigned, there will we a 2 week washout period, then return to clinic for light assignment then light exposure for 10 week, similar visits as described below.

For the follow up clinic visit or phone call (Week 10), data similar to the information gathered at the initial visit will be collected. The description of the pain (burning, electrical, shooting…etc.) and its location will be reviewed. A physical examination assessing for pain and sensation to light touch that is part of the standard of care will be provided for the participants. At the end of the study, the participants will be asked to return the LED strip, their logs and questionnaires.

There is an optional blood draw and saliva sample collection for patients that consent to this. Blood and saliva samples will be collected at baseline and end of study, blood draws will be done to look for inflammatory mediators, increased anti inflammatory mediators and endocannabinoids. Saliva samples will be collected to check for melatonin.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 - 80 able to understand English and comply with study protocol
* Peripheral neuropathy from HIV or chemotherapy.
* History of fibromyalgia
* Headaches
* Chronic Pain
* 7-day average numeric pain score of 5/10 or greater at baseline evaluation

Exclusion Criteria:

* Subjects receiving remuneration for their pain treatment
* Subjects that are incarcerated
* Subjects unable to read English and complete assessments
* Addictive behavior, severe clinical depression, or psychotic features

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mohab Ibrahim, PhD., MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center South, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] Hooley JM, Franklin JC, Nock MK. Chronic pain and suicide: understanding the association. Curr Pain Headache Rep. 2014;18(8):435. doi: 10.1007/s11916-014-0435-2. PMID 24916035
- [Background] Hassett AL, Aquino JK, Ilgen MA. The risk of suicide mortality in chronic pain patients. Curr Pain Headache Rep. 2014;18(8):436. doi: 10.1007/s11916-014-0436-1. PMID 24952608
- [Result] Smith AA, Friedemann ML. Perceived family dynamics of persons with chronic pain. J Adv Nurs. 1999 Sep;30(3):543-51. doi: 10.1046/j.1365-2648.1999.01123.x. PMID 10499210
- [Result] Gray D, Coon H, McGlade E, Callor WB, Byrd J, Viskochil J, Bakian A, Yurgelun-Todd D, Grey T, McMahon WM. Comparative analysis of suicide, accidental, and undetermined cause of death classification. Suicide Life Threat Behav. 2014 Jun;44(3):304-16. doi: 10.1111/sltb.12079. PMID 25057525
- [Result] Hwang MH, Shin JH, Kim KS, Yoo CM, Jo GE, Kim JH, Choi H. Low level light therapy modulates inflammatory mediators secreted by human annulus fibrosus cells during intervertebral disc degeneration in vitro. Photochem Photobiol. 2015 Mar-Apr;91(2):403-10. doi: 10.1111/php.12415. Epub 2015 Jan 26. PMID 25557915
- [Derived] Martin L, Porreca F, Mata EI, Salloum M, Goel V, Gunnala P, Killgore WDS, Jain S, Jones-MacFarland FN, Khanna R, Patwardhan A, Ibrahim MM. Green Light Exposure Improves Pain and Quality of Life in Fibromyalgia Patients: A Preliminary One-Way Crossover Clinical Trial. Pain Med. 2021 Feb 4;22(1):118-130. doi: 10.1093/pm/pnaa329. PMID 33155057
- [Derived] Martin LF, Patwardhan AM, Jain SV, Salloum MM, Freeman J, Khanna R, Gannala P, Goel V, Jones-MacFarland FN, Killgore WD, Porreca F, Ibrahim MM. Evaluation of green light exposure on headache frequency and quality of life in migraine patients: A preliminary one-way cross-over clinical trial. Cephalalgia. 2021 Feb;41(2):135-147. doi: 10.1177/0333102420956711. Epub 2020 Sep 9. PMID 32903062

RESULTS

PARTICIPANT FLOW:
Groups:
- Exposure to White LED Light Crossed Over to Green LED.: Subjects will exposed to white light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks
  Exposure to white LED light: Participants will be exposed to white LED strip lights in a dark room for 2 hours a day.
Period: Overall Study
Arm/Group | Exposure to White LED Light Crossed Over to Green LED.
Started | 55
Completed | 53
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Exposure to White LED Light and Crossover to Green LED Light.: Subjects will exposed to white light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks
  Exposure to white LED light: Participants will be exposed to white LED strip lights in a dark room for 2 hours a day.
  Subjects will exposed to green light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks.
  Exposure to green LED light: Participants will be exposed to green LED strip lights in a dark room for 2 hours a day.
  Subject will be exposed to white light (sham) for 10 weeks, then have a wash out period for 2 weeks, then exposed to green light (experimental) for 10 weeks.
  Exposure to green LED light: Participants will be exposed to green LED strip lights in a dark room for 2 hours a day.
  Exposure to white LED light: Participants will be exposed to white LED strip lights in a dark room for 2 hours a day.
Arm/Group | Exposure to White LED Light and Crossover to Green LED Light.
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: For Chronic Pain
Description: Change in the intensity of chronic pain as measured by the Numerical Pain Scale (NPS). The NPS has a value ranging from 0 to 10 out of a maximum of 10. 0 means no pain. 10 means the most severe pain.
Time Frame: baseline and 10 - 22 weeks, depending on study arm
Population: Adult patients with chronic pain
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Exposure to White LED Light: Subjects will be exposed to white light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks
- Green LED Light Exposure: Subjects will be exposed to green light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks
Arm/Group | Exposure to White LED Light | Green LED Light Exposure
Number analyzed (Participants) | 55 | 55
score on a scale | 0.45 (0.2) | 3.7 (0.4)

2. Secondary Outcome: Fibromyalgia Impact Questionnaire
Description: Change in Fibromyalgia Impact Questionnaire (FIQ) total score. The FIQ is a validated, self-reported measure assessing physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being over the past week. Scores range from 0 to 100, with higher scores indicating greater impairment.
Time Frame: baseline and 10 - 22 weeks, depending on study arm
Population: patients with fibromyalgia
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Green Light Exposure: Fibromyalgia patients exposed to green LED light
Arm/Group | Exposure to White LED Light | Green Light Exposure
Number analyzed (Participants) | 55 | 55
score on a scale | 10.43 (3.46) | 28.92 (4.32)

3. Secondary Outcome: Headache Impact Test-6
Description: Change in Headache Impact Test-6 (HIT-6) total score from baseline to 10-22 weeks. The HIT-6 is a 6-item questionnaire designed to assess the impact of headaches on daily life, including pain severity, disability, and emotional effects over the past 4 weeks. Scores range from 36 to 78, where 36-49 indicates little or no impact, 50-55 indicates some impact, 56-59 reflects substantial impact, and 60-78 indicates severe impact requiring intervention. A higher score indicates greater headache impact.
Time Frame: baseline and 10 - 22 weeks, depending on study arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure to White LED Light | Exposure to Green LED Light
Number analyzed (Participants) | 55 | 55
score on a scale | 1.14 (1.3) | 12.85 (1.6)

4. Secondary Outcome: EQ-5D-5L
Description: Change in health-related quality of life as measured by the EQ-5D-5L. The EQ-5D-5L is a standardized, patient-reported outcome measure that assesses health-related quality of life across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on a 5-level scale (no problems to extreme problems). The score is calculated using a country-specific value set to produce a single index value ranging from -0.594 (worse than death) to 1.0 (perfect health), where higher scores indicate better health status.
Time Frame: baseline and 10 - 22 weeks, depending on study arm
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Green Light Exposure: Exposure to green LED light: Participants will be exposed to green LED strip lights in a dark room for 2 hours a day.
Arm/Group | Exposure to White LED Light | Green Light Exposure
Number analyzed (Participants) | 55 | 55
score on a scale | 0.13 (0.03) | 0.28 (0.04)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 22 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov definitions.
Groups:
- Exposure to Green LED Light: Subjects will be exposed to green light provided to them, in their homes in a dark room for approximately 2 hours for 10 weeks
Arm/Group | Exposure to White LED Light | Exposure to Green LED Light
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT03677206/Prot_000.pdf
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03677206/ICF_001.pdf